CLINICAL TRIAL: NCT01523275
Title: A Randomized Study of Mitomycin-C Application in the Endoscopic Surgical Treatment of Patients With Laryngotracheal Stenosis
Brief Title: Study of Mitomycin-C Application in Laryngotracheal Stenosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to poor patient accrual, the study was closed prior to reaching the desired study size
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Laryngotracheal Stenosis
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-04

CONDITIONS: Laryngeal Stenosis; Subglottic Stenosis; Tracheal Stenosis
Keywords: mitomycin-C; laryngotracheal stenosis; subglottic stenosis; tracheal stenosis; endoscopic airway surgery
MeSH Terms: conditions — Laryngostenosis; Tracheal Stenosis | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mitomycin-C (Experimental): Patients will undergo standard endoscopic surgical treatment for LTS involving CO2 laser radial incisions and balloon dilation, as well as topical application of MMC in the radial incisions.
  Interventions: Drug: Mitomycin -C
- Saline (Placebo Comparator): Patients will undergo standard endoscopic surgical treatment for LTS involving CO2 laser radial incisions and balloon dilation, as well as topical application of isotonic saline in the radial incisions.
  Interventions: Other: Saline application

INTERVENTIONS:
Drug: Mitomycin -C — Topical mitomycin-C at a dosage of 0.4mg/ml will be applied to cottonoid pledgets and placed into the radial incisions for 3 minutes.
  Arms: Mitomycin-C
Other: Saline application — Isotonic saline will be applied to cottonoid pledgets and placed into the patient's radial incisions for 3 minutes as the placebo intervention.
  Arms: Saline

SUMMARY:
This is a randomized, prospective, double-blind, placebo-controlled clinical trial of the use of mitomycin-C topical application as an adjunctive treatment in the endoscopic surgical treatment of patients with laryngotracheal stenosis. We hypothesize that the use of mitomycin-C improves patient outcome in the endoscopic surgical treatment of laryngotracheal stenosis.

DETAILED DESCRIPTION:
Obstruction of the upper airway caused by laryngotracheal stenosis (LTS) often results in severe morbidity and even mortality. Treatment of LTS continues to present a challenge and a wide array of surgical techniques have been employed. Despite multiple endoscopic and/or open reconstructive procedures, patients often experience restenosis as a result of the abnormal wound-healing process that initially instigated the airway obstruction. The high rate of stenosis relapse has therefore motivated researchers to find new methods to modulate and control the wound-healing process of the airway. Although other adjuvant treatments such as steroids and antibiotics have been investigated in LTS, much attention in recent years has turned to the use of topical mitomycin-C (MMC). As a topical application, MMC has been shown to inhibit fibroblast proliferation in wound-healing processes. The use of MMC in the treatment of airway stenosis was first reported in 1998 and is now routinely used in the endoscopic management of LTS. However, despite numerous animal and human studies, the benefit of MMC in LTS patients remains questionable. While previously published retrospective data suggest that the addition of MMC improves outcome, there have been no prospective studies to directly address the efficacy of MMC in endoscopic LTS surgery. This study will be the first randomized, prospective, double-blind, placebo controlled clinical trial designed to investigate the efficacy of MMC as an adjunctive therapy to endoscopic surgical treatment in patients with LTS. In addition, the study will investigate the relationship between patient symptoms and objective pulmonary function measurements. Ultimately, the results of this study may influence the treatment and evaluation of patients with laryngotracheal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with laryngotracheal stenosis, including subglottic stenosis or tracheal stenosis
* Patients with disease amenable to treatment with endoscopic CO2 laser radial incisions and balloon dilation
* Age greater than or equal to 18 years

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Patients with glottic and supraglottic stenosis
* Patients with disease not amenable to treatment with endoscopic CO2 laser radial incisions and balloon dilation
* Patients with cartilaginous subglottic or tracheal stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Yung, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF - Voice and Swallowing Clinic, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from the UCSF Voice and Swallowing Center clinic from August 1, 2012 to February 1, 2018
Groups:
- Mitomycin C: Endoscopic dilation with topical mitomycin C
- Saline: Endoscopic dilation with topical saline
Period: Overall Study
Arm/Group | Mitomycin C | Saline
Started | 6 | 9
Completed | 4 | 7
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Mitomycin-C | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years of age] | 57.1 (12.4) | 48 (8.3) | 53 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 8 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Age of Onset [Mean (Standard Deviation); unit: Years] — Mean age of participants when they had onset of laryngotracheal stenosis
  Years | 52.2 (13.5) | 44.2 (9.2) | 49 (12.3)
Etiology [Count of Participants; unit: Participants]
  Idiopathic | 6 | 5 | 11
  Granulomatosis with Polyangiitis | 2 | 1 | 3
  Post-Intubation | 1 | 0 | 1
Site [Count of Participants; unit: Participants]
  Subglottis | 8 | 5 | 13
  Trachea | 1 | 0 | 1
  Subglottis and Trachea | 0 | 1 | 1
Prior laryngotracheal stenosis surgery [Count of Participants; unit: Participants]
  Yes | 4 | 5 | 9
  No | 5 | 1 | 6
Average prior laryngotracheal stenosis surgeries [Mean (Standard Deviation); unit: Surgeries] | 1.1 (1.5) | 4 (4.9) | 2 (3.5)
Prior treatment with Mitomycin C [Count of Participants; unit: Participants]
  Yes | 3 | 4 | 7
  No | 6 | 2 | 8
Prior treatment with Kenalog [Count of Participants; unit: Participants]
  Yes | 2 | 4 | 6
  No | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time to Repeat Surgery
Description: Length of time between surgeries for laryngotracheal stenosis during the study
Time Frame: 24 months
Population: Patients who did not undergo a subsequent surgery after the initial study surgery were excluded as a surgical interval could not be calculated. There were two patients in each arm that did not have subsequent surgeries
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Saline | Mitomycin-C
Number analyzed (Participants) | 7 | 4
Months | 17.9 (15.7) | 17.4 (12.8)
Statistical Analysis 1: Comparison: Saline vs Mitomycin-C; Test type: Equivalence — Analysis of 44 subjects (22 in each arm) would provide 90% power to detect a difference in the time interval to reoperation of 6 months between the two treatment arms, at an alpha level of 0.05. This difference of 6 months is clinically meaningful and is smaller than previous case series studies would suggest. However, due to poor patient accrual, the study was closed prior to reaching the desired study size; p = 0.95, t-test, 2 sided

2. Secondary Outcome: Duration of Symptom Improvement
Description: Symptom improvement was measured using the Clinical COPD Questionnaire, a 10-point patient reported symptom score. Duration of symptom improvement was defined as the time from surgery to the time that symptoms to worsened beyond a CCQ score of 1 or the time to the subsequent surgery if CCQ never exceeded 1
Time Frame: 24 months
Population: Time to symptom score (CCQ) progression was calculated for each surgery performed during the study with available CCQ data.
Measure: Mean (Standard Deviation); unit: Months
Units Other Than Participants: Surgeries
Arm/Group | Saline | Mitomycin-C
Number analyzed (Participants) | 9 | 6
Number analyzed (Surgeries) | 13 | 9
Months | 4.1 (6.7) | 6.0 (6.4)
Statistical Analysis 1: Comparison: Saline vs Mitomycin-C; Test type: Equivalence — A difference of 6 months to symptom progression is clinically meaningful; p = 0.52, t-test, 2 sided

3. Secondary Outcome: Peak Inspiratory Flow Measurement
Description: Change in maximum inspiratory air flow from preoperative value to highest postoperative value within 3 months of surgery. Calculation details: Highest postoperative value within 3 months of surgery minus preoperative value.
Time Frame: 3 months
Population: Improvement in peak inspiratory flow (PIF) was calculated for each surgery performed during the study with available PIF data
Measure: Mean (Standard Deviation); unit: Liters per second
Units Other Than Participants: Surgeries
Arm/Group | Saline | Mitomycin-C
Number analyzed (Participants) | 9 | 6
Number analyzed (Surgeries) | 14 | 8
Liters per second | 1.1 (1.5) | 1.3 (0.96)
Statistical Analysis 1: Comparison: Saline vs Mitomycin-C; Test type: Equivalence — 0.5 liters per second is clinically significant; p = 0.64, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through study completion, which was on average of 2.3 years
Arm/Group | Saline | Mitomycin-C
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT01523275/Prot_SAP_000.pdf